CLINICAL TRIAL: NCT06631131
Title: Evaluation of the Dentoskeletal Effects of Maxillary Molar Distalization With Clear Aligners: Class II Elastic Anchorage vs. Miniscrew Anchorage
Brief Title: Distalization With Aligners: Anchorage Options
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 40173
Record Dates: First submitted 2024-09-27; First posted 2024-10-08 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Class II Malocclusion; Class II Malocclusion, Division 1
Keywords: Class II malocclusion; Clear aligners; Distalization; Miniscrew anchorage
MeSH Terms: conditions — Overbite; Malocclusion, Angle Class II

STUDY DESIGN:
Intervention Model Description: A total of twenty-seven patients were initially included. However, five patients were excluded because they discontinued treatment (n=2), had poor treatment compliance (n=2), or had poor radiograph quality (n=1). Consequently, the final sample comprised 22 individuals, with 11 individuals (22 second molar, 22 first molar and 22 second premolar) in each group, ranging in age from 15 to 25. All patients were treated with clear aligners.The patients were divided into two groups, those who were treated with sequential distalization with aligners supported by Class II elastics (group 1) or IZC miniscrews (group 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Distalization with clear aligners supported by Class II elastics (Active Comparator): Group 1: these patients were treated with sequential distalization with aligners supported by Class II elastics.
  Interventions: Device: Distalization with clear aligners supported by Class II elastics
- Distalization with clear aligners supported by miniscrew (Active Comparator): Group 2: these patients were treated with sequential distalization with aligners supported by IZC miniscrews.
  Interventions: Device: Distalization with clear aligners supported by miniscrew

INTERVENTIONS:
Device: Distalization with clear aligners supported by Class II elastics — Sequential distalization (50%) with clear aligners was planned in the maxillary arch for each patient. ). In group 1, with the beginning of the movement of the upper first molars, Class II intermaxillary elastics were used from precision cuts of the upper canines to the buttons on the lower first molars for supporting distalization movement.
  Arms: Distalization with clear aligners supported by Class II elastics
Device: Distalization with clear aligners supported by miniscrew — Sequential distalization (50%) with clear aligners was planned in the maxillary arch for each patient. In group 2, IZC miniscrews were inserted in the IZC region between the upper molars in both sides before first molar movement started. The same intramaxillary elastics were used from precision cuts of the upper canines to the IZC miniscrew for supporting distalization movement.
  Arms: Distalization with clear aligners supported by miniscrew

SUMMARY:
Background: To compare the dentoskeletal effects of Class II elastic anchorage and infrazygomatic crest (IZC) miniscrew anchorage in sequential maxillary molar distalization using clear aligners.

Methods: A total of 22 patients with Angle Class II malocclusion treated with clear aligners and maxillary molar distalization were included. Based on the anchorage method patients were divided into two groups: Class II elastics (Group 1) or IZC miniscrews (Group 2). Lateral cephalometric radiographs and digital models were obtained from all patients before treatment (T0) and after distalization of the second premolars (T1) to assess skeletal and dental changes. Geomagic Control X was used to superimpose the digital models.

DETAILED DESCRIPTION:
The data for this study were obtained from patients who presented for treatment at the Department of Orthodontics at Bezmialem Vakif University Faculty of Dentistry. All patients were treated with clear aligners (Invisalign®, Align Technology, CA, USA) at Bezmialem University Hospital. Sequential distalization (50%) was planned in the maxillary arch. For each aligner, a staging of 0.25 mm was determined. Distalization starts with the second molars, then the first molars after half of the second molar movement is completed, and finally the premolars. In the ClinCheck planning, 3 or 4 mm vertical rectangular attachments were placed from the second molar to the canine and were bevelled mesially to enhance the distalization forces. The patients were divided into two groups, those who were treated with sequential distalization with aligners supported by Class II elastics (group 1) or IZC miniscrews (group 2). In group 1, with the beginning of the movement of the upper first molars, Class II intermaxillary elastics were used from precision cuts of the upper canines to the buttons on the lower first molars. In group 2, IZC miniscrews were inserted in the IZC region between the upper molars in both sides before first molar movement started. The same intramaxillary elastics were used from precision cuts of the upper canines to the IZC miniscrew. The use of intra/intermaxillary elastics was started with the initiation of upper first molar movement to prevent anchorage loss and maxillary incisor proclination. Both groups were instructed to wear the elastics and aligners a minimum of 22 hours per day using a 10-day aligner wear protocol. Maxillary third molars were extracted before treatment.

Patients were scanned by iTero 5D Element intraoral scanner and radiographs were taken before treatment (T0) and after distalization of the second premolar (T1).

Cephalometric radiographs were obtained from all patients and these radiographs were used for two-dimensional measurements.Digital tracing and measurements of the cephalometric radiographs were performed using NemoCeph version 6.0 software. Angular dental measurements were performed between the long axis of the teeth and the sella-nasion (S-N) plane using Image J software. The long axis was determined as a line through the incisal edge and the root apex for the incisors, through the buccal cusp tip and the root apex for the premolars, and through the centroid and the furcation for the molars. Digital models were exported from OrthoCAD software as stereolithography (STL) files and imported into Geomagic Control X software for three-dimensional (3D) model comparison. All digital models were superimposed using the local best fit algorithm. A reference area in the palatal region was used for the model superimposition and 50 iteration points were defined in this area for the superimpositions.

After model superimposition, reference points of the teeth were selected on the two models to enable linear measurements. These points were the mesiobuccal cusp tips of the maxillary molars and the buccal cusp tips of the premolars. These reference points were marked on the T0 and T1 models and measurements were taken to observe changes on all three axis. In linear measurements,

1. X-axis represent buccolingual (transversal) differences (X+ in the buccal direction and X- in the palatal direction);
2. Y-axis represent mesiodistal (sagittal) differences (Y+ in the distal direction and Y- in the mesial direction); and
3. Z-axis represent vertical differences (Z+ indicating extrusion and Z- indicating intrusion).

For angular measurements, reference points and vectors were identified on 3D models. These points were the mesiobuccal and mesiopalatal cusp tips of the molars and the buccal and palatal cusp tips of the premolars. The angles between reference vectors were measured. Rotational movements were measured using the XY-axis, with positive values indicating mesiobuccal rotation and negative values indicating distobuccal rotation.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were as follows:

1. Class II molar relationship,
2. mild or moderate dental crowding on both arches,
3. previous extraction or absence of the upper third molars,
4. good compliance to orthodontic treatment,
5. availability of initial and progress stereothography (STL) files of intraoral scans and lateral cephalometric radiographs.

Exclusion Criteria:

Exclusion criteria were

1. severe dental crowding on both arches,
2. Class II subdivision malocclusion,
3. severe skeletal Class II malocclusion requiring orthognathic surgery,
4. presence of impacted or supernumerary teeth,
5. tooth extraction (except third molars),
6. poor compliance to orthodontic treatment,
7. craniofacial and dentofacial disorders, syndromes, or systemic diseases impacting bone metabolism or tooth movement.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Dentoskeletal Effects of Maxillary Molar Distalization with Clear Aligners: Class II Elastic Anchorage vs. Miniscrew Anchorage | Patients were collected and treatmets were started up to 9 months. At 12 weeks, miniscrews were inserted in group 2 and elastics were started to be used in each group. Final data were collected up to 20 months.
  Lateral cephalometric radiographs and digital models were obtained from all patients before treatment and after distalization of the second premolars to assess skeletal and dental changes.
  Digital tracing and measurements of the cephalometric radiographs were performed by the same investigator using NemoCeph software. Angular dental measurements were performed between the long axis of the teeth and the sella-nasion (S-N) plane using Image J software.
  Geomagic Control X was used to superimpose the digital models and measurement of dental movements.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Sunal Aktürk, Assistant professor, Study Director — University of Health Sciences, Hamidiye Faculty of Dental Medicine, Department of Orthodontics; Ezgi Kösen, PhD student, Principal Investigator — Bezmialem Vakif University,Institute of Health Sciences, Department of Orthodontics,
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data of this study belong to the PhD thesis and the thesis has not yet been defended.